CLINICAL TRIAL: NCT06235554
Title: Feasibility Study Evaluating the Safety and Efficacy of the Renal Stimulation by Direct Wire Pacing, During Renal Denervation Procedure.
Acronym: RNS by DWP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ceric Sàrl (Industry)
Collaborators: Electroducer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A01789-36
Record Dates: First submitted 2024-01-11; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Essential Hypertension
Keywords: Renal Stimulation; Renal Denervation procedure
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Intervention Model Description: Feasibility study, prospective, open-label, single center, single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental)
  Interventions: Procedure: Renal Stimulation

INTERVENTIONS:
Procedure: Renal Stimulation — Renal Denervation procedure as per hospital routine practice
  Other Names: Renal Dernervation

SUMMARY:
The goal of this feasibility study is to evaluate the safety and efficacy of the Renal Stimulation (RNS) by Direct Wire Pacing, during Renal Denervation (RDN) procedure in patient candidate for renal denervation with the ParadiseTM System. The main questions it aims to answer are:

* Is the RNS before RDN a straightforward method, allowing quantification of the renal sympathetic traffic?
* Does the RNS increase blood pressure (SBP), and is this increase significantly blunted after RDN?
* Does the 3-month 24h SBP decrease correlated with the RNS-induced SBP change before RDN?
* Can the difference between RNS-induced SBP rise before and after RDN be used as a procedural endpoint for RDN? Participants will be asked for their agreement to conduct an RNS before and after the RDN. No additional experimental procedure will be added to the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing and able to comply with the protocol and has provided written informed consent.
* Age ≥18
* Patient candidate for renal denervation with the ParadiseTM System based on physician's assessment.
* Patients affiliated to a social security system

Exclusion Criteria:

* Patients who meet any of the contraindications listed in the Instructions for Use of ParadiseTM Ultrasound Renal Denervation System will be excluded:

  * Renal arteries diameter < 3 mm and > 8 mm
  * Patient with relevant renal artery disease (% diameter stenosis > 30%, aneurysm or fibromuscular disease)
  * Stented renal artery
  * Iliac/femoral artery stenosis precluding insertion of the ParadiseTM catheter
  * Known allergy to contrast medium
* Patient with known secondary cause of hypertension
* Patient with contraindication to chronic anticoagulation therapy or heparin
* Patient with Type 1 diabetes mellitus
* Patient with more than one accessory renal artery
* Woman currently pregnant or breastfeeding
* Patient with other concomitant conditions that may adversely affect the patient or the study outcome
* Patient with mental or physical inability to participate in the study
* Patient under judicial protection, tutorship, or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of occurrence of adverse events | Three month after procedure
  safety of the renal nerves stimulation performed by Direct Wire Pacing technique during renal denervation procedure
efficacy on Systolic Blood Pressure change to be measured with a blood pressure monitor | Three month after procedure
  efficacy of the renal nerves stimulation performed by Direct Wire Pacing technique during renal denervation procedure

SECONDARY OUTCOMES:
Impact on Systolic Blood Pressure | Three month after procedure
  Investigate the impact of the renal denervation in the Renal Nerves Stimulation induced Systolic Blood Pressure change.
Systolic Blood Pressure as response prediction tool | Three month after procedure
  Investigate whether Renal Nerves Stimulation induced Systolic Blood Pressure change before Renal Denervation could be a reliable tool to predict mid-term Renal Denervation response
Systolic Blood Pressure variation as response prediction tool | Three month after procedure
  Investigate whether difference in Renal Nerves Stimulation-induced Systolic Blood Pressure change before and after Renal Denervation could be a reliable tool to predict mid-term Renal Denervation